CLINICAL TRIAL: NCT06316843
Title: A Randomized, Double-Blinded, Placebo-Controlled, Pilot Study of the Combination of Valacyclovir + Celecoxib (IMC-2) for the Treatment of Post-Acute Sequelae of SARS-CoV-2 Infection in Adults
Brief Title: Valacyclovir Plus Celecoxib for Post-Acute Sequelae of SARS-CoV-2
Acronym: PASC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bateman Horne Center (Other)
Responsible Party: Principal Investigator, LUCINDA BATEMAN, MD, Medical Director, Bateman Horne Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BHC202 v2.1
Record Dates: First submitted 2024-03-11; First posted 2024-03-19 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2024-10

CONDITIONS: Long COVID; PASC Post Acute Sequelae of COVID 19
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome | interventions — DMAC2L protein, human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- 1500 Valacyclovir 200 Celecoxib (Experimental): Treatment will consist of four blue 375mg valacyclovir capsules and one white 200 mg celecoxib capsule
  Interventions: Drug: Valacyclovir celecoxib dose 1
- 750 Valacyclovir 200 Celecoxib (Experimental): Treatment will consist of two blue 375mg valacyclovir capsules, two blue placebo capsules, and one white 200 mg celecoxib capsule
  Interventions: Drug: Valacyclovir celecoxib dose 2
- Matched Color Placebo Capsules (Placebo Comparator): Treatment will consist of four blue placebo capsules and one white placebo capsule
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Valacyclovir celecoxib dose 1 — 1500 mg valacyclovir 200 mg celecoxib taken two times a day
  Other Names: Arm 1
  Arms: 1500 Valacyclovir 200 Celecoxib
Drug: Valacyclovir celecoxib dose 2 — 750 mg valacyclovir 200 celecoxib mg taken two times a day
  Other Names: Arm 2
  Arms: 750 Valacyclovir 200 Celecoxib
Drug: Placebo — Placebo capsules colored matched to investigational product taken two times a day
  Other Names: Arm 3
  Arms: Matched Color Placebo Capsules

SUMMARY:
To explore the safety and efficacy of daily doses of celecoxib + valacyclovir in the treatment of patients with prolonged symptoms caused by COVID-19.

DETAILED DESCRIPTION:
This is a randomized, double-blinded, placebo-controlled, single-center, three arm, 12-week study designed to explore the safety and efficacy of daily doses of valacyclovir + celecoxib for the treatment of prolonged symptoms caused by COVID-19 infection in adult female patients. The treatment consists of twice daily doses of valacyclovir and celecoxib, which is theorized to provide potent suppression of tissue-resident herpes viruses subsequently activated by an initial infection with the SARS-CoV-2 virus. The physiological response to tissue-resident herpes virus activation is in turn hypothesized to be causally related to symptoms associated with the Post-Acute Sequelae of SARS-CoV-2 Infection (PASC). There are three arms and in each arm, patients take four blue capsules and one white capsule in the morning and again in the evening. The capsules dispensed for arm 1 will consist of four 375mg valacyclovir capsules and one 200 mg celecoxib capsule. Arm 2 will be dispensed two blue 375mg valacyclovir capsules, two blue placebo capsules and one white 200 mg celecoxib capsule. Arm 3 will be dispensed four blue placebo capsules and one white placebo capsule.

Approximately 60 female patients will be enrolled at Bateman Horne Center for this study.

Candidates will undergo initial pre-screening by telephone or database review, after which, if they appear to meet initial entry criteria, they will have an in- person screening visit. They will start recording symptom data, starting at the baseline visit, and continuing with weekly recordings, for the duration of their study participation. Each week, the patient will provide information on their average fatigue, sleep quality and pain intensity.

Patients with underlying medical or psychiatric conditions that could impact their safe participation in the study or interfere with their ability to complete or comply with the study's requirements will not be enrolled. In addition, any patient dependent upon opioids/narcotics (collectively referred to as "opioids") for pain control for any reason will not be enrolled in the study.

Due to the celecoxib component of the combination therapy, patients using NSAIDs or COX-2 inhibitors will need to discontinue use of NSAIDs at least 7 days before randomization. NSAIDs including PRN usage should not be utilized for the duration of the study. Instead, acetaminophen may be utilized as needed throughout the study (but not to exceed 3250 mg per day). Patients may also continue low-dose aspirin for cardioprotection (< 325 mg/day).

Patients may remain on stable doses of SSRIs and other non-excluded anti- depressants; however, poorly controlled, or severely depressed patients should not be enrolled. Only clinically stable and well-controlled patients should be considered, i.e., patients with mild to moderate depression who in the judgement of the investigator are not at risk of suicidal ideation or behavior.

For all patients a screening visit will be conducted so the PI or Sub-I can ensure that all entry criteria have been satisfied. At baseline, the PI/sub-I will ensure all safety laboratory results are satisfactory, any required washout has been completed and all entry criteria have been met. Patients should initiate study drug treatment on the day of the Baseline visit (Day 1), followed by BID dosing for the duration of the study.

Blood and urine will be collected at the Screening visit for safety assessments. Urine pregnancy tests will be performed at Week 4, 8 and 12 (or early termination) visits for patients with child-bearing potential. A blood sample for safety labs will be collected during Week 12/ET. Urine drug screening for drugs of abuse will be conducted at the Screening visit; patients positive for cocaine, methamphetamine, phencyclidine (PCP), methadone, non-disclosed amphetamines and non-disclosed opiates will be screen failed. Patients positive for disclosed, prescribed opioids at the Screening visit, yet deemed suitable for washout, must be able to remain off all opioids for the duration of the study and have a negative repeat UDS at the Baseline visit. Additional drug testing may be conducted at the PI or Sub-I's discretion.

Patients with clinically significant renal insufficiency or a history of renal disease (as defined in the entry criteria) will be excluded.

Patients will have in-person study visits scheduled for Screening, Baseline, Weeks 4, 8 and 12/ET. If necessary, remote visits may be substituted for the Week 4 and/or Week 8 visits. A follow-up survey or phone call will be scheduled approximately 2 weeks after completion of study drug treatment at Week 12 or ET.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to read, understand, and sign the informed consent.
2. Female at birth, 18-65 years of age at the time of study entry.
3. Must have smartphone with internet access to complete surveys online.
4. Diagnosis of Long COVID according to any of the following definitions Infected individuals will have a history of suspected, probable, or confirmed SARS-CoV-2 infection as defined by WHO criteria and at least three months of persistent fatigue and muscle weakness, functional impairment, and cognitive impairment since the acute infection.

Adults with suspected SARS-CoV-2 infection. An adult qualifies as having suspected SARS-CoV-2 infection if meeting at least one of the following criteria (a-e) below:

a. Clinical criteria: Acute onset of fever and cough OR acute onset of any three or more of the following signs or symptoms: fever, cough, general weakness /fatigue, headache, myalgia, sore throat, coryza, dyspnea, anorexia/nausea/vomiting, diarrhea, altered mental status. These patients should also meet one of the following epidemiological criteria: i. Epidemiological criteria:

1. Residing or working in an area with a high risk of transmission of virus: closed residential settings, humanitarian settings such as camp and camp-like settings for displaced persons; anytime within the 14 days before symptom onset; or
2. Residing or travel to an area with community transmission anytime within the 14 days before symptom onset; or
3. Working in any health care setting, including within health facilities or the community, anytime within the 14 days before symptom onset.

   b. A patient with severe acute respiratory illness: (acute respiratory infection with history of fever or measured fever of ≥38C°; and cough; with onset within the last ten days; and requires hospitalization).

   c. An asymptomatic patient not meeting any of the epidemiologic criteria above but with a previously positive SARS-CoV-2 Antigen- RDT.

   d. Adults with probable SARS-CoV-2 infection. An adult qualifies as having probable SARS-CoV-2 infection if meeting any one of 1-3 below: i. A patient who meets clinical criteria for suspected SARS- CoV-2 AND is a contact of a probable or confirmed case or linked to a COVID-19 cluster; ii. A suspect case with chest imaging showing findings suggestive of COVID-19 disease; iii. A person with recent onset of anosmia (loss of smell) or ageusia (loss of taste) in the absence of any other identified cause; e. Adults with confirmed SARS-CoV-2 infection. An adult qualifies as having confirmed SARS-CoV-2 infection if meeting any one of 1-4 below: i. Any person with a positive Nucleic Acid Amplification Test (NAAT); ii. Any person with of a positive SARS-CoV-2 Antigen-RDT AND meeting either the probable case definition or suspect criteria A OR B; iii. An asymptomatic person with a positive SARS-CoV-2 Antigen-RDT who is a contact of a probable or confirmed case; iv. Any person with a positive SARS-CoV-2 nucleocapsid protein antibody test OR a positive SARS-CoV-2 spike protein antibody test IF not vaccinated

5. Women of child-bearing potential must have a negative serum pregnancy test at screening and agree to on-site urine pregnancy testing at all subsequent study visits. Women confirmed to be of non-childbearing potential do not require pregnancy testing. Pregnancy tests will not be required for remote visits. To be considered of non-child-bearing potential, the patient must be:

a. Post-menopausal (defined as no menses for at least one year); or b. Surgically sterile (s/p hysterectomy, bilateral oophorectomy, or bilateral tubal ligation at least six months prior to beginning treatment with study drug); or c. At least three months s/p a non-surgical permanent sterilization procedure 6. A urine drug screen performed at the Screening Visit must be negative for drugs of abuse such as methamphetamine, cocaine, phencyclidine (PCP), and non-disclosed amphetamines and opioids/opiates. The following stipulations also apply:

1. Patients with a positive screening UDS due to prescribed amphetamines for allowed conditions do not require further UDS testing. They may proceed with study treatment, assuming no evidence of abuse or dependency.
2. Patients positive for prescribed opioids at the Screening Visit yet deemed appropriate for washout and study participants must have a negative repeat UDS at the Baseline Visit.

   7. Patients must be willing and able to withdraw and refrain from chronic use of antivirals (as defined in Exclusion Criterion, below). In the judgement of the investigator, it must be medically advisable for these therapies to be withdrawn.

   8. Qualified patients with mild to moderate depression who in the judgment of the investigator are not at risk of suicidal ideation or behavior. The dose of allowed antidepressants should have been stable for at least 30 days prior to Baseline Visit..

   9. In the opinion of the Investigator, the patient is willing and able to comply with all protocol-specified requirements.

   10. Women of child-bearing potential must be willing to utilize an effective birth control method for the duration of the study. Allowable contraceptive methods include:

a. Oral, implantable, injectable, or transdermal hormonal contraceptives (should have been used for a minimum of one full cycle prior to administration of study drug) b. Intrauterine devices (IUD) c. Double barrier method (male or female condom, sponge, diaphragm, or vaginal ring with simultaneous use of spermicidal jelly or cream) 11. Patients should not require routine treatment with warfarin, heparin, lithium, digoxin, amiodarone, isoniazid, phenytoin, fluconazole, methotrexate, probenecid, or raloxifene. Patients on these medications should not be screened. PRN usage of fluconazole for short time periods is permitted.

12. Patients must have successfully completed at least two PROMIS Fatigue and two PROMIS Sleep Disturbance surveys a minimum of 7 days apart during the interval leading up to the baseline visit.

Exclusion Criteria:

1. Breastfeeding, pregnant, or planning to become pregnant during the next six months.
2. In the opinion of the Investigator, any clinically significant, uncontrolled, or unstable medical or surgical condition that could affect the patient's ability to participate in the study or potentially compromise her well-being while enrolled in the study.
3. In the opinion of the Investigator or based on results of the HADS, evidence of a clinically significant psychiatric disorder; e.g., severe, unstable or poorly controlled depression, anxiety or obsessive-compulsive disorder; moderate or severe alcohol use disorder; substance use disorder other than mild cannabis use disorder; or any history of bipolar disorder, schizophrenia, schizoaffective disorder or other psychotic disorder.
4. A score of >15 on the Patient Health Questionnaire-9 (PHQ-9) determined by survey at screening.
5. A positive response to thoughts of suicide or self-harm on the PHQ-9 determined by survey at screening.
6. A diagnosis of ME/CFS prior to January 2020.
7. Any anticipated need for surgery that in the opinion of the Principal Investigator or Sub-I might confound results or interfere with the patient's ability to comply with the protocol.
8. Symptomatic and/or otherwise clinically significant cardiac disease, including but not limited to myocardial infarction during the preceding two years; uncontrolled hypertension; symptomatic heart failure (e.g., New York Heart Association Class II or higher); angina or other evidence of significant coronary artery disease; clinically significant cardiac rhythm or conduction abnormality or anticipation of bypass or other cardiac surgery within the next 12 months.
9. Acute non-COVID systemic infection (e.g., HIV, hepatitis) or other active viral or bacterial infection during the screening/washout period or at the Baseline visit. (Patient may remain in screening until the active infection has resolved, or re-screen after recuperation.)
10. Currently receiving chronic systemic corticosteroids (>5 mg prednisone daily, or equivalent).
11. Uncontrolled sleep apnea. Patients successfully treated with CPAP or other devices are eligible.
12. Use of chronic nucleoside analog antiviral suppression therapy within one month of the Screening Visit or requiring on average more than one acute treatment course every two months.
13. Current use of celecoxib either alone or in combination with valacyclovir or famciclovir
14. In the opinion of the Investigator, evidence of current drug or alcohol abuse or dependency, or history of abuse or dependence during the preceding 12 months.
15. The patient has undergone a malabsorptive weight loss procedure (e.g., Roux-en-Y or other bypass procedure).
16. Severe IBS-C or colonic inertia as evidenced by seven or more days between bowel movements.
17. History of significant adverse reaction or allergy to sulfonamides, celecoxib, famciclovir, acyclovir, valacyclovir or penciclovir cream (Denavir®).
18. History of aspirin-sensitive asthma, or any other history of other allergic- type reactions after taking aspirin or other NSAID such as asthma or urticaria.
19. History of Sulfa Allergy.
20. History of peptic ulcer disease or upper gastrointestinal bleeding that is thought to pose a significant risk of GI bleeding with the daily use of celecoxib.
21. Clinically significant elevations of AST, ALT, or bilirubin at the screening assessment (or at the last assessment prior to baseline, if repeated) in the opinion of the Investigator.
22. Presence of active kidney disease, as evidenced by an estimated glomerular filtration rate (eGFR) of less than 60 mL/min/1.73m2.
23. History of acute kidney injury within the past year, any history of chronic kidney disease stage 3 or higher.
24. In the opinion of the Investigator, evidence of other clinically significant laboratory abnormality(ies) based on the screening laboratory assessments and/or medical history.
25. Untreated, symptomatic gall bladder disease (i.e., symptoms within preceding six months).
26. Plans to undergo vaccination against Herpes varicella/ zoster (i.e., shingles or chickenpox) during the study. Instead, vaccination should be completed at least 14 days prior to the Baseline Visit or delayed until at least two weeks after the last dose of study medication.
27. Patients known or suspected to be slow CYP2C9 metabolizers based on genotype or previous history/experience with other CYP2C9 substrates (such as warfarin, phenytoin, glimepiride, tolbutamide, celecoxib, meloxicam, piroxicam, or ibuprofen).
28. Investigational drug usage within 30 days of Screening.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2023-10-15 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Fatigue assessed with the Patient-Reported Outcomes Measurement Information System (PROMIS) Fatigue 7a Instrument | 12 weeks
  The PROMIS Fatigue 7a will be automatically calculated to a T-score with a standard error of 4. Higher fatigue T-scores represent worse than average fatigue. The primary efficacy analysis will be the mean change from baseline (MCFB) to Week 12 in fatigue based on the weekly survey PROMIS Fatigue 7a T-scores. A mixed models for repeated measures (MMRM) procedure will be used to compare the MCFB between the treatment and placebo arm.

CONTACTS AND LOCATIONS:
Overall Officials: Lucinda Bateman, MD, Principal Investigator — Bateman Horne Center
Locations (1):
- Bateman Horne Center, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No